CLINICAL TRIAL: NCT02754882
Title: A Phase 3, Randomised, Double-blind Study to Compare the Efficacy, Safety, PK and Immunogenicity Between SB8 (Proposed Bevacizumab Biosimilar) and Avastin® in Subjects With Metastatic or Recurrent Non-squamous Non-small Cell Lung Cancer
Brief Title: A Study Comparing SB8 and Avastin® in Patients With Advanced Non-squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB8-G31-NSCLC
Record Dates: First submitted 2016-03-24; First posted 2016-04-28 (Estimated); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: NSCLC; bevacizumab; avastin
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab (Avastin) (Active Comparator): Avastin® + Carboplatin/Paclitaxel
  Interventions: Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- SB8 (A proposed bevacizumab biosimilar) (Experimental): SB8 + Carboplatin/Paclitaxel
  Interventions: Drug: SB8; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Bevacizumab — Avastin® 15 mg/kg IV every 3 weeks on Day 1
  Other Names: Avastin®
  Arms: Bevacizumab (Avastin)
Drug: SB8 — SB8 15 mg/kg IV every 3 weeks on Day 1
  Other Names: SB8 (A proposed bevacizumab biosimilar)
  Arms: SB8 (A proposed bevacizumab biosimilar)
Drug: Carboplatin — Carboplatin AUC 6 IV every 3 weeks on Day 1 for 4-6 cycles
Drug: Paclitaxel — Paclitaxel 200 mg/m2 IV every 3 weeks on Day 1 for 4-6 cycles
  Other Names: Taxol

SUMMARY:
This study is designed to establish biosimilarity of SB8, a proposed biosimilar product of bevacizumab, to EU-sourced bevacizumab, in patients with metastatic or recurrent non-squamous non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Standard efficacy parameters, safety profiles, pharmacokinetics and immunogenicity will be compared between SB8 and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. ECOG performance status of 0-1
3. Histologically-confirmed metastatic or recurrent non-squamous non-small cell lung cancer
4. At least one measurable lesion according to RECIST v1.1.
5. Able to receive bevacizumab, carboplatin and paclitaxel based on adequate laboratory and clinical parameters

Exclusion Criteria:

1. Diagnosis of small cell carcinoma of the lung or squamous cell carcinoma
2. Sensitizing EGFR mutations or ALK rearrangements
3. Increased risk of bleeding determined by investigator based on radiographic / clinical findings
4. History of systemic chemotherapy administered in the first-line setting for metastatic or recurrent disease of NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 763 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Reck, M.D., Principal Investigator — LungenClinic Grosshansdorf, Germany
Locations (104):
- Belarus (6):
  - Brest Regional Oncology Dispensary, Brest
  - Grodno Regional Clinical Hospital, Grodno
  - N. N. Alexandrov Republican Scientific and Practical Center of Oncology and Medical Radiology, Lesnoy
  - Minsk city Clinical Oncological Dispensary, Minsk
  - Mogilev Regional Oncological Dispensary, Mogilev
  - Vitebsk Regional Clinical Oncological Dispensary, Vitebsk
- Georgia (8):
  - JSC Maritime Hospital, Batumi
  - JSC Saint Nikolozi Surgery Center, Kutaisi
  - LTD Research Institute of Clinical Medicine, Tbilisi
  - ICO-Institute of Clinical Oncology, Tbilisi
  - New Vision University Hospital, Tbilisi
  - LTD MediClubGeorgia, Tbilisi
  - Institute for Personalized Medicine LTD, Tbilisi
  - LTD Chemotherapy and Immunotherapy Clinic Medulla, Tbilisi
- Germany (8):
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - University Hospital Homburg, Homburg
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Leipzig [Pneumologie], Leipzig
  - Klinik Löwenstein, Löwenstein
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
- Hungary (6):
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - Orszagos Koranyi Tbc Es Pulmonologiai Intezet, Iv. Tudobel, Budapest
  - Csongrád Megyei Önkormányzat Mellkasi Betegségek Szakkó, Deszk
  - Veszprem Megyei Onkormanyzat Tudogyogyintezete, Farkasgyepű
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz - Rendeloint, Szolnok
  - Markusovszky Egyetemi Oktatókórház, Szombathely
- Poland (3):
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
  - MED-POLONIA Sp.z o.o., Poznan
- Romania (11):
  - Med Life, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Medisprof, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Constanta, Constanța
  - Centrul de Oncologie Sf. Nectarie, Craiova
  - Oncolab, Craiova
  - Radiotherapy Center CJ radioterapie si chimioterapie adulti, Floreşti
  - Centrul de Oncologie Euroclinic, Iași
  - Institutul Regional de Oncologie Iasi, Iași
  - Pelican Impex, Oradea
  - Oncocenter Oncologie Clinica, Timișoara
- Russia (21):
  - State Budgetary Institution of Arkhangelsk Oblast "Arkhangelsk Region Clinical Oncology Center, Arkhangelsk
  - State Budgetary Healthcare Institution "Chelyabinsk Regional Clinical Oncology Center", Chelyabinsk
  - State Autonomous Healthcare Institution "Republican Clinical Oncology Center of Ministry of Healthcare of Tatarstan Republic", Kazan'
  - State Budgetary Healthcare Institution "Regional Clinical Hospital #1 n.a. professor S.V. Ochapovsky" of Ministry of Healthcare of Krasnodar Region, Krasnodar
  - Federal State Budgetary Scientific Institution " N.N. Blokhin Russian Cancer Research Center" of the Ministry of Health of the Russian Federation, Moscow
  - State Autonomous Healthcare Institution of Moscow "Moscow City Oncology Hospital # 62 of Healthcare Department of Moscow", Moscow
  - State Regional Budgetary Healthcare Institution "Murmansk Regional Oncology Center", Murmansk
  - State Budgetary Healthcare Institution of Nizhny Novgorod oblast "Nizhny Novgorod Region Oncology Center", Nizhny Novgorod
  - State Budgetary Healthcare Institution of Novosibirsk Region "Novosibirsk Region Clinical Oncology Center", Novosibirsk
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncology Center", Omsk
  - Federal Budgetary Healthcare Insittution "Saint-Petersburg Clinical Hospital of RAS", Saint Petersburg
  - State Budgetary Healthcare Institution Leningradskaya Region Clinical Hospital, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education "Academician I.P. Pavlov First St. Petersburg State Medical University" of the Ministry of Healthcare of the Russian Federation./ Scientific Research Institute of Pulmonology, Saint Petersburg
  - Federal State Budgetary Institution " Scientific Research Institute of Oncology n.a. N.N. Petrov" of Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Clinical Oncology Center", Saint Petersburg
  - Private foundation of Educational establishment of Higher Education Medical University "REAVIZ", Samara
  - State Budgetary Healthcare Institution " Oncology Center #2" of Krasnodar Region Ministry of Healthcare, Sochi
  - State Budgetary Healthcare Institution Republican Clinical Oncology Center of Ministry of Healthcare of the Republic of Bashkortostan, Ufa
  - State Budgetary Healthcare Institution "Volgograd Regional Clinical Oncology Center", Volzhskiy
  - State Budgetary Healthcare Institution of Yaroslavl Region "Regional Clinical Oncology Hospital", Yaroslavl
  - State Budgetary Healthcare Institution of Sverdlovskaya Oblast "Sverdlovsk Regional Oncology Center", Yekaterinburg
- Serbia (4):
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Center Kragujevac, Clinic for Pulmology, Kragujevac
  - Clinical Centre Nis, Niš
- South Korea (10):
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - CHA Bundang Medical Center, CHA University, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Yonsei Universtiy, Wonju Severance Christian Hospital, Wŏnju
- Spain (9):
  - C.H. Provincial de Castellón, Castellon
  - H.U. Severo Ochoa, Leganés
  - H.G.U. G. Marañón, Madrid
  - H.U. F. Jiménez Díaz, Madrid
  - C.H. de Orense, Ourense
  - Clínica Universidad de Navarra, Pamplona
  - H.U. Sant Joan de Reus, Reus
  - C.H.U. de Canarias, Santa Cruz de Tenerife
  - H.U.N. Sra. Valme, Seville
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chang Gung Medical Foundation, Linkou, Taoyuan District
- Thailand (5):
  - Siriraj Hospital, Bangkok
  - ChiangMai Univerisity, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Prince of Songkla University, Hat Yai
  - Udonthani Cancer Hospital, Udon Thani
- Ukraine (8):
  - Komunalna ustanova "Chernivetskyi oblasnyi klinichnyi onkolo, Chernivtsi
  - Komunalnyi zaklad Miska bahatoprofilna klinichna likarnia #4, Dnipropetrovsk
  - Kharkivskyi oblasnyi onkologichnyi klinichnyi tsentr, Kharkiv
  - Khmelnytskyi oblasnyi onkolohichnyi dyspanser, Khmelnytskyi
  - Odeskyi oblasnyi onkolohichnyi dyspanser, Odesa
  - OKZ "Sumskyi oblasnyi klinichnyi onkolohichnyi dyspanser", Sumy
  - Vinnytskyi oblasnyi klinichnyi onkolohichnyi dyspanser, Vinnytsia
  - Zaporozhye Regional Clinical Oncology Center, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab (Avastin) | SB8 (A Proposed Bevacizumab Biosimilar)
Started | 384 | 379
Completed | 38 | 35
Not Completed | 346 | 344

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab (Avastin) | SB8 (A Proposed Bevacizumab Biosimilar) | Total
Number analyzed (Participants) | 384 | 379 | 763
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 269 | 255 | 524
  >=65 years | 115 | 124 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.18) | 60.2 (8.95) | 60.1 (20.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 127 | 255
  Male | 256 | 252 | 508
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 35 | 32 | 67
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 348 | 347 | 695
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.49 (4.707) | 25.50 (4.809) | 25.50 (4.755)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Overall Response (Best Overall Response Rate[ORR]) by 24 Weeks
Description: The best ORR was defined as the proportion of subjects whose best overall response was either Complete Response (CR) or Partial Response (PR) according to RECIST v1.1 during the induction treatment period by 24 weeks.
  CR: Disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 24 weeks from randomisation
Population: The Full Analysis Set consisted of all randomised subjects. The subjects were analysed based on the treatment they were randomised to by intention-to-treat principle. However, subjects who did not qualify for randomisation and were inadvertently randomised into the study were excluded from FAS, provided these subjects did not receive any IP, and there was one subject who met these criteria. So, there is a difference between "Started" in Participant Flow module and Analysis Population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab (Avastin) | SB8 (A Proposed Bevacizumab Biosimilar)
Number analyzed (Participants) | 383 | 379
percentage of participants | 42.8 | 47.6
Statistical Analysis 1: Comparison: Bevacizumab (Avastin) vs SB8 (A Proposed Bevacizumab Biosimilar); Test type: Equivalence — Pre-defined equivalence margin was [0.737, 1.357]; Risk Ratio (RR) = 1.11, 90% CI 2-sided [0.975 to 1.269] — SB8 vs. Avastin

2. Secondary Outcome: Progression Free Survival
Description: PFS is defined as the time from the date of Randomisation to the date of disease progression (progressive disease [PD]) or death regardless of the cause of death.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: from the date of randomisation to the date of disease progression or death up to 12 months from randomisation of the last subject
Population: Full Analysis Set (FAS): Consisted of all randomised subjects. The subjects were analysed based on the treatment they were randomised to by intention-to-treat principle. Per-protocol Set (PPS): Consisted of all FAS subjects who completed at least first 2 cycles of combination chemotherapy with a tumour assessment and did not have any major protocol deviations that impacted the primary efficacy assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 379 | 383
months
  FAS | 8.50 [7.40 to 9.70] | 7.90 [7.40 to 9.50]
  PPS: number analyzed (Participants) | 337 | 328
  PPS | 8.50 [7.20 to 9.70] | 7.90 [7.30 to 9.40]

3. Secondary Outcome: Overall Survival
Description: OS was defined as the time from the date of randomisation to the date of death regardless of the cause of death.
  Subjects who were alive at the time of analysis were censored at the date of last known alive.
Time Frame: from the date of randomisation to the date of death up to 12 months from randomisation of the last subject
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 379 | 383
months
  FAS | 14.90 [13.30 to 17.10] | 15.80 [13.60 to 17.10]
  PPS: number analyzed (Participants) | 337 | 328
  PPS | 14.80 [13.00 to 17.10] | 15.80 [13.80 to 17.70]

4. Secondary Outcome: Duration of Response (DoR)
Description: DoR in subjects with response from documented tumour response until disease progression up to 12 months from randomisation of the last subject
Time Frame: from documented tumour response until disease progression up to 12 months from randomisation of the last subject
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: months
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 379 | 383
months
  FAS | 6.38 (3.773) | 6.79 (4.117)
  PPS: number analyzed (Participants) | 337 | 328
  PPS | 6.33 (3.784) | 6.81 (4.177)

5. Secondary Outcome: Number of Participants With Treatment-related Adverse Events Using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03
Description: After the end of treatment (EOT) visit, SAEs should be reported to the Sponsor if the Investigator becomes aware of them.
  Severity Grade of NCI-CTCAE v4.03 Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) (Instrumental ADL refers to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.) Grade 3: Severe or medically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation indicated; disabling; limiting self-care ADL (Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.) Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death related to AE
Time Frame: AEs were reported from the time the informed consent form (ICF) was signed until the EOT visit, approximately 24 months from study initiation.
Population: Safety Set (SAF): The Safety Set consisted of all subjects who received the study drug at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 378 | 380
Participants
  TEAEs | 348 | 346
  CTCAE Grade 1 | 47 | 57
  CTCAE Grade 2 | 127 | 134
  CTCAE Grade 3 | 119 | 97
  CTCAE Grade 4 | 33 | 31
  CTCAE Grade 5 | 22 | 27

6. Secondary Outcome: Pharmacokinetics: Trough Level [Ctrough]
Description: Ctrough at selected cycles (i.e., Cycle 1, 3, 5 and 7)
Time Frame: Up to 21 weeks (Cycle 1,3,5 and 7. Each cycle is 21 days.)
Population: Pharmacokinetic Population (PK Population): This set consisted of subjects allocated to PK sub-study who had at least one measured serum concentration of bevacizumab.
  PK analyses were performed on the PK population. The number of participants analyzed in each Cycle is the number of participants in PK population with non-missing values or without protocol deviation for PK blood sampling at the cycle.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 161 | 180
ug/mL
  Cycle 1: number analyzed (Participants) | 142 | 166
  Cycle 1 | 0.0000 (0.00000) | 0.0000 (0.00000)
  Cycle 3: number analyzed (Participants) | 137 | 152
  Cycle 3 | 83.7568 (44.49701) | 102.3939 (69.36822)
  Cycle 5: number analyzed (Participants) | 118 | 141
  Cycle 5 | 109.0906 (50.65915) | 119.9343 (54.65786)
  Cycle 7: number analyzed (Participants) | 100 | 121
  Cycle 7 | 121.7382 (62.62150) | 133.7669 (58.84136)

7. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration [Cmax]
Description: Maximum Plasma Concentration (Cmax) at selected cycles (i.e., Cycle 1, 3, 5 and 7)
Time Frame: Up to 21 weeks (Cycle 1,3,5 and 7. Each cycle is 21 days.)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 161 | 180
ug/mL
  Cycle 1: number analyzed (Participants) | 155 | 170
  Cycle 1 | 306.0352 (98.71872) | 302.6362 (87.10467)
  Cycle 3: number analyzed (Participants) | 133 | 146
  Cycle 3 | 374.9657 (106.54366) | 399.4598 (136.27431)
  Cycle 5: number analyzed (Participants) | 114 | 140
  Cycle 5 | 389.3132 (123.07791) | 397.6183 (125.84175)
  Cycle 7: number analyzed (Participants) | 98 | 119
  Cycle 7 | 397.5435 (120.74092) | 426.1350 (144.24538)

8. Secondary Outcome: Immunogenicity Assessments (Anti-drug Antibodies)
Description: Incidence of anti-drug (bevacizumab) antibodies (ADA)
  The incidence of overall ADA results (i.e. Positive, Negative, Inconclusive) was presented by treatment group at Cycle 7 and the end of treatment (EOT). Overall ADA result was defined as below:
  * 'Positive' for a subject with treatment-induced or treatment-boosted ADA, where treatment-induced ADA indicated at least one positive result after pre-dose of Cycle 1 for subjects with negative ADA at pre-dose of Cycle 1, and treatment-boosted ADA indicated at least one positive result with higher titre level compared to pre-dose of Cycle 1 after pre-dose of Cycle 1 for subjects with positive ADA at pre-dose of Cycle 1.
  * 'Negative' for a subject without positive ADA until Cycle 7 and EOT.
  * 'Inconclusive' for a subject with positive ADA at Cycle 1 and without positive result with higher titre level observed after pre-dose of Cycle 1 up to Cycle 7 and EOT.
Time Frame: Up to 21 weeks (Cycle 1,3,5, 7 and EOT visit. Each cycle is 21 days.), approximately 24 months from study initiation.
Population: The analysis was performed using the Safety Set (SAF). The SAF consisted of all subjects who received the study drug at least once. This analysis set was used for the safety analyses. The subjects were analysed based on the treatment they received.
  There were 4 subjects in Avastin group and 1 subject in SB8 group who had not received any IP or non-IP treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 378 | 380
Participants
  Cycle 1 (BL): number analyzed (Participants) | 372 | 371
  Cycle 1 (BL): Positive | 15 | 15
  Cycle 1 (BL): Negative | 357 | 356
  Cycle 1 (BL): Inconclusive (only applicable for "Overall") | 0 | 0
  Cycle 3: number analyzed (Participants) | 338 | 338
  Cycle 3: Positive | 29 | 22
  Cycle 3: Negative | 309 | 316
  Cycle 3: Inconclusive (only applicable for "Overall") | 0 | 0
  Cycle 5: number analyzed (Participants) | 301 | 296
  Cycle 5: Positive | 15 | 21
  Cycle 5: Negative | 286 | 275
  Cycle 5: Inconclusive (only applicable for "Overall") | 0 | 0
  Cycle 7: number analyzed (Participants) | 266 | 279
  Cycle 7: Positive | 28 | 20
  Cycle 7: Negative | 238 | 259
  Cycle 7: Inconclusive (only applicable for "Overall") | 0 | 0
  EOT: number analyzed (Participants) | 150 | 161
  EOT: Positive | 21 | 9
  EOT: Negative | 129 | 152
  EOT: Inconclusive (only applicable for "Overall") | 0 | 0
  Cycle 7 Overall: number analyzed (Participants) | 341 | 337
  Cycle 7 Overall: Positive | 46 | 34
  Cycle 7 Overall: Negative | 284 | 294
  Cycle 7 Overall: Inconclusive (only applicable for "Overall") | 11 | 9
  EOT Overall: number analyzed (Participants) | 341 | 337
  EOT Overall: Positive | 55 | 37
  EOT Overall: Negative | 276 | 291
  EOT Overall: Inconclusive (only applicable for "Overall") | 10 | 9

9. Secondary Outcome: Immunogenicity Assessments (Neutralizing Antibodies)
Description: Incidence of anti-drug (bevacizumab) antibodies (ADA) - neutralizing antibodies (NAb) The analysis was performed using the Safety Set (SAF). Overall Number of Participants Analyzed represents the number of subjects in SAF.
  The total number is not the sum of the number of subjects of each visits, since NAb results only for subjects with ADA positive against SB8 or Avastin were used for the summary.
  Number Analyzed of each visit is equal to the number of subjects with ADA positive of each visit, which is displayed in 8. Secondary Outcome: Immunogenicity Assessments (Anti-drug Antibodies).
Time Frame: Up to 21 weeks (Cycle 1,3,5, 7 and EOT visit. Each cycle is 21 days.), approximately 24 months from study initiation.
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 378 | 380
Participants
  Cycle 1 (BL): number analyzed (Participants) | 15 | 15
  Cycle 1 (BL): Positive | 0 | 1
  Cycle 1 (BL): Negative | 15 | 14
  Cycle 3: number analyzed (Participants) | 29 | 22
  Cycle 3: Positive | 9 | 9
  Cycle 3: Negative | 20 | 13
  Cycle 5: number analyzed (Participants) | 15 | 21
  Cycle 5: Positive | 5 | 8
  Cycle 5: Negative | 10 | 13
  Cycle 7: number analyzed (Participants) | 28 | 20
  Cycle 7: Positive | 12 | 11
  Cycle 7: Negative | 16 | 9
  EOT: number analyzed (Participants) | 21 | 9
  EOT: Positive | 9 | 5
  EOT: Negative | 12 | 4

10. Other Pre Specified Outcome: Best Objective Response Rate by 11 and 17 Weeks
Description: Best Objective Response Rate (ORR) by 11 weeks and 17 weeks
Time Frame: 11 weeks and 17 weeks from randomisation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SB8 (A Proposed Bevacizumab Biosimilar) | Bevacizumab (Avastin)
Number analyzed (Participants) | 379 | 383
Participants
  11 Weeks (FAS) | 107 | 100
  11 Weeks (PPS): number analyzed (Participants) | 337 | 328
  11 Weeks (PPS) | 99 | 89
  17 Weeks (FAS) | 159 | 152
  17 Weeks (PPS): number analyzed (Participants) | 337 | 328
  17 Weeks (PPS) | 149 | 137

ADVERSE EVENTS:
Time Frame: AEs were reported from the time the ICF was signed until the EOT visit, approximately 24 months from study initiation.
Description: All safety analyses were performed using the Safety Set (SAF). The SAF consisted of all subjects who received the study drug at least once. This analysis set was used for the safety analyses. The subjects were analysed based on the treatment they received.
  There were 4 subjects in Avastin group and 1 subject in SB8 group who had not received any IP or non-IP treatment.
Arm/Group | Bevacizumab (Avastin) | SB8 (A Proposed Bevacizumab Biosimilar)
All-Cause Mortality (participants affected / at risk) | 171/380 | 166/378
Serious Adverse Events (participants affected / at risk) | 81/380 | 75/378
Other Adverse Events (participants affected / at risk) | 316/380 | 323/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (Avastin) (N=380) | SB8 (A Proposed Bevacizumab Biosimilar) (N=378)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 6 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (7) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Optic atrophy (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Sudden death (General disorders) | 6 (6) | 4 (4)
Infusion site extravasation (General disorders) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 7 (8)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis glandularis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2)
Internal haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (Avastin) (N=380) | SB8 (A Proposed Bevacizumab Biosimilar) (N=378)
Anaemia (Blood and lymphatic system disorders) | 87 (107) | 87 (102)
Neutropenia (Blood and lymphatic system disorders) | 69 (119) | 74 (122)
Thrombocytopenia (Blood and lymphatic system disorders) | 45 (68) | 57 (96)
Leukopenia (Blood and lymphatic system disorders) | 23 (44) | 39 (59)
Nausea (Gastrointestinal disorders) | 79 (224) | 74 (177)
Diarrhoea (Gastrointestinal disorders) | 24 (26) | 29 (38)
Vomiting (Gastrointestinal disorders) | 20 (23) | 24 (32)
Constipation (Gastrointestinal disorders) | 18 (24) | 20 (24)
Asthenia (General disorders) | 43 (55) | 49 (58)
Fatigue (General disorders) | 46 (58) | 46 (56)
Weight decreased (Investigations) | 28 (30) | 37 (37)
Aspartate aminotransferase increased (Investigations) | 24 (38) | 32 (48)
Alanine aminotransferase increased (Investigations) | 30 (42) | 29 (47)
Blood urea increased (Investigations) | 18 (37) | 28 (50)
Blood alkaline phosphatase increased (Investigations) | 27 (34) | 26 (36)
Decreased appetite (Metabolism and nutrition disorders) | 34 (47) | 36 (39)
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 (92) | 46 (117)
Myalgia (Musculoskeletal and connective tissue disorders) | 35 (57) | 24 (37)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (31) | 19 (55)
Neuropathy peripheral (Nervous system disorders) | 54 (59) | 38 (39)
Paraesthesia (Nervous system disorders) | 32 (34) | 32 (33)
Headache (Nervous system disorders) | 27 (49) | 26 (29)
Peripheral sensory neuropathy (Nervous system disorders) | 35 (36) | 24 (25)
Proteinuria (Renal and urinary disorders) | 24 (40) | 17 (25)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 24 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (21) | 23 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (31) | 21 (21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 20 (28)
Alopecia (Skin and subcutaneous tissue disorders) | 183 (184) | 184 (185)
Hypertension (Vascular disorders) | 35 (45) | 46 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT02754882/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT02754882/SAP_001.pdf